CLINICAL TRIAL: NCT04506619
Title: Long-Term Safety and Efficacy Outcomes Following Previously Administered Short-Term Treatment With SHP607 in Extremely Premature Infants
Brief Title: Safety and Efficacy Outcomes Following Previously Administered Short-Term Treatment With SHP607 in Extremely Premature Infants
Status: Terminated | Type: Observational
Why Stopped: As the revised OHB-607-202 protocol extends the study's observational arm through 24 months corrective age (CA), the SHP607-203 protocol was terminated at 24 months CA.
Sponsor: Oak Hill Bio Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: SHP607-203; 2020-002726-84 (EudraCT Number)
Record Dates: First submitted 2020-07-27; First posted 2020-08-10 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2022-04

CONDITIONS: Retinopathy of Prematurity (ROP); Intraventricular Hemorrhage; Bronchopulmonary Dysplasia; Chronic Lung Disease of Prematurity
MeSH Terms: conditions — Retinopathy of Prematurity; Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- SHP607 250 mcg/kg/24 hours: Participants who received 250 micrograms per kilogram per 24 hours (mcg/kg/24 hours) in the previous study SHP607-202 (NCT03253263) will be followed into this long-term study SHP607-203.
  Interventions: Other: No Intervention
- SHP607 400 mcg/kg/24 hours: Participants who received 400 mcg/kg/24 hours in the previous study SHP607-202 (NCT03253263) will be followed into this long-term study SHP607-203.
  Interventions: Other: No Intervention
- Standard Neonatal Care: Participants who received standard neonatal care in the previous study SHP607-202 (NCT03253263) will be followed into this long-term study SHP607-203.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This is a non-interventional study.

SUMMARY:
The purpose of this study is to evaluate long-term safety and efficacy outcomes following previously administered short-term exposure to SHP607, as compared to a standard neonatal care group.

DETAILED DESCRIPTION:
In this long-term follow-up study, participants who enrolled in SHP607-202 (NCT03253263) will be followed from 12 months corrected age (CA) through 60 months CA. Participants will not receive any investigational product in this study.

ELIGIBILITY:
Inclusion Criteria:

* Participants who were randomized into Study SHP607-202 (NCT03253263). Participants who were randomized, but did not complete Study SHP607-202 (NCT03253263) must be at least 12 months CA.
* Written informed consents (and assents, if applicable) must be signed and dated by the participant's parent(s)/legally authorized representative(s) prior to any study-related procedures. The informed consent and any assents for underage parents must be approved by the institutional review board (IRB)/independent ethics committee (IEC).

Exclusion Criteria:

- Participants are excluded from the study if the participant or participant's parent(s)/legally authorized representative(s) is/are unable to comply with the protocol or is/are unlikely to be available for long-term follow-up as determined by the investigator.

Ages: 12 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants who previously received SHP607 or standard neonatal care in Study SHP607-202 (NCT03253263) are planned to be enrolled in Study SHP607-203.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-08-05 (Actual)

PRIMARY OUTCOMES:
Number of Emergency Room Visits | 12 months CA through 60 months CA
  Number of emergency room visits associated with a respiratory diagnosis will be reported.
Number of Hospitalizations | 12 months CA through 60 months CA
  Number of hospitalizations associated with a respiratory diagnosis will be reported.
Incidence of Signs and Symptoms of Respiratory Disease | 12 months CA through 60 months CA
  Incidence of signs and symptoms of respiratory disease (yes/no) is assessed by recording episodes of wheezing, coughing, and respiratory medication.
Number of Days of Respiratory Medication Use | 12 months CA through 60 months CA
  Number of days of respiratory medication use (for example, bronchodilators, steroids, leukotriene inhibitors, diuretics) will be reported.
Total Number of Days on Home Respiratory Technology use | 12 months CA through 60 months CA
  Total number of days on home respiratory technology use (for example, home oxygen, continuous positive airway pressure [CPAP], tracheostomy) will be reported.
Number of Participants With Adverse Events (AEs) | 12 months CA through 60 months CA
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Growth Parameters: Body Weight | At 12, 24, and 60 months CA
  Body weight is measured in kilograms (kg) without shoes and with light clothing using a calibrated scale.
Growth Parameters: Body Length | At 12 and 24 months CA
  Body length is a supine measurement from the top of the head to the sole of the foot with the participant lying on the back with hips and knees extended.
Growth Parameters: Height | At 60 months CA
  Height is a measure of participant from head to foot (standing measure). A stadiometer should be utilized for measurement of height.
Growth parameters: Head circumference | At 12 and 24 months CA
  Head circumference or occipital frontal circumference is measured over the occiput and just above the supraorbital ridge, which is the largest circumference of the head.
Physical Development as Assessed by Physical Examination | At 12, 24, and 60 months CA
  Physical examinations will include a review of the participant's general appearance.
Physical Development as Assessed by Neurological Examination for Assessment of Cerebral Palsy | At 12, 24, and 60 months CA
  Neurological examination for the diagnosis of cerebral palsy (CP) will be conducted. Neurologic examinations for the diagnosis of CP will be conducted by physicians including assessment of motor function, strength and development, muscle tone, and postural and movement abnormalities.
Physical Development as Assessed by Visual Acuity | At 12, 24, and 60 months CA
  Visual acuity is a measure of how well a participant sees at different distances. It will be categorized as the following: normal (measurable acuity greater than or equal to [>=] 20/40); below normal (20/200 less than or equal to [<=] measurable acuity <20/40); poor (measurable acuity <=20/200); blind/low vision (only the ability to detect the 2.2 centimeter [cm] wide stripes on the low-vision Teller acuity card and at any location in the visual field).
Cognitive Development Assessed by Bayley Scales of Infant and Toddler Development (BSID-III) | At 24 months CA
  The BSID-III will be used to assess cognitive, motor, and language skills, and is applicable to children aged 1-42 months. The BSID-III is an assessment tool designed to measure a young child's skills in the 3 core areas of development: cognitive, language, and motor. There are 5 subscales, the cognitive subscale (Score range: 55-145) stands alone while the 2 language subscales (expressive and receptive) combine to make a total language score (Range: 47-153) and the 2 motor subtests (fine and gross motor) form a combined motor scale (Range: 46-154). A positive value indicates improvement.
Cognitive Development Quotient Assessed by Kyoto Scale of Psychological Development (KSPD) | At 24 months CA
  KSPD is a alternative scale to the BSID and used to assess cognitive, motor, and language skills at Japan sites only. The KSPD is a validated neurodevelopmental outcome assessment that is standardized for Japanese children and has been evaluated in comparison to BSID in the assessment of developmental characteristics of very low birth weight Japanese infants. The KSPD is designed to measure a young child's skills in three domains of development: Cognitive-Adaptive (non-verbal reasoning or visuospatial perception), Language-Social (interpersonal relationships, socialization, verbal abilities), and Postural-Motor (fine and gross motor functions). The scale consists of 328 items covering a Cognitive-Adaptive area, Language-Social area, and Postural-Motor area. For each of the three areas, a sum score is converted to a Developmental Quotient (dividing the developmental age by the chronological age and then multiplying the quotient by 100). A positive value indicates improvement.
Cognitive Development Assessed by Wechsler Preschool and Primary Scale of Intelligence (WPPSI) | At 60 months CA
  The WPPSI is a measure of general cognitive development in children that has components of both verbal and non-verbal tasks. It is applicable to preschoolers and young children aged 2 years +6 months to 7 years +7 months, and is a direct assessment of a child's cognitive skills. The standard score For the WPPSI ranges from Below 70 (extremely low) to above 130 (very superior).
Gross Motor Function Assessed by Gross Motor Function Measure-88 (GMFM-88) | At 24 and 60 months CA
  The GMFM-88 item scores is used to calculate a domain-specific percent score for each of the 5 GMFM-88 dimensions, which are the following: Lying and rolling; Sitting; Crawling and kneeling; Standing; Walking, running, and jumping. Each of the 88 items is rated on a 4-point scale: 0=does not initiate; 1=initiates; 2=partially completes; and 3=completes. The GMFM-88 total scores range from 0% (no mobility) to a score of 100%. The test is considered to be appropriate for children whose motor skills are at or below those of a 5-year-old child without any motor disability. The GMFM-88 will be administered at 24 months CA. GMFM-88 Sections D (Standing) and E (Walking, Running and Jumping) only will be administered at 5 years CA.
Childhood Behavior Assessed by Vineland Adaptive Behavior Scales (VABS-III) | At 24 and 60 months CA
  The VABS-III test measures adaptive behaviors, including the ability to cope with environmental changes, to learn new everyday skills, and to demonstrate independence. This test measures the following 4 key domains: communication, daily living skills, socialization, and motor skills. The score ranges from 20 to 140 on which higher scores indicate a higher level of better behavior.
Childhood Behavior Assessed by Attention-Deficit/Hyperactivity Disorder Rating Scale (ADHD-RS-V) | At 60 months CA
  The ADHD-RS-V measures the behaviors of children with Attention-Deficit/Hyperactivity Disorder (ADHD). It consists of 18 items designed to reflect current symptomatology of ADHD based on DSM-V criteria. Each item is scored from a range of 0 (reflecting no symptoms) to 3 (reflecting severe symptoms) with total scores ranging from 0-54. The 18 items are grouped into 2 subscales: hyperactivity-impulsivity (even numbered items 2-18) and inattention ("inattentiveness") (odd numbered items 1-17).
Childhood Behavior Assessed by Social Communication Questionnaire (SCQ) | At 60 months CA
  The SCQ is a brief instrument that helps evaluate communication skills and social functioning in children that can be used for screening for autism or autism spectrum disorders (ASD) in the general population. The score ranges from 0 to 39, with a cut off of greater than (>) 15 indicating ASD.
Health Related Quality of Life (HRQoL) Assessed by the Pediatric Quality of Life Inventory (PedsQL) Scales | At 24, 36, 48, and 60 months CA
  HRQoL will be assessed via the validated Pediatric Quality of Life Inventory (PedsQL) Scales appropriate for the child's age of development. The following scales will be used in this study: Infant Scale for ages 13-24 months (45 Items); Toddler Scale for 2-4 years of age (21 Items); Young Child Scale for 5-7 years of age (23 Items). Scores are transformed to a 0 to 100 scale. Higher scores indicate better quality of life.
Health Status Measured by the Health Utilities Index 2/3 | At 60 months CA
  The Health Utilities Index (HUI) is a family of generic health profiles and preference-based systems used for measuring health status, reporting HRQoL, and producing utility scores. The HUI 2/3 system contains a number of attributes/domains to classify the level of health status. Each attribute or domain (eg, mobility, cognition, emotion or pain) is rated on a 5-point ordinal scale to indicate the severity level, ranging from 1-5 (higher numbers indicating a more severe level).
Healthcare Resource Utilization | 12 months CA through 60 months CA
  Healthcare resource utilization is measured by the number of in-patient and outpatient visits, including emergency room visits and visits to specialists.
Number of Participants With Targeted Medical Events and Fatal Serious Adverse Events (SAEs) | 12 months CA through 60 months CA
  Targeted medical events are intracranial hypertension, any abnormality of glucose metabolism (eg, hypoglycemia, hyperglycemia, and diabetes), tonsillar hypertrophy (based on tonsil examination [part of the physical examination]), and increased cardiac size. A serious adverse event (SAE) is defined as an untoward medical occurrence that at any dose meets one or more of the following criteria: outcome is fatal/results in death, is life-threatening, requires inpatient hospitalization or results in prolongation of an existing hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect, is a medically important event.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (3):
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Robert Wood Johnson Medical School, New Brunswick, New Jersey
- Italy (3):
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Istituto G Gaslini Ospedale Pediatrico IRCCS - INCIPIT - PIN, Genova
  - Presidio Ospedaliero Di Treviso Ca' Foncello, Treviso
- Ashford and St. Peter's Hospitals NHS Trust - St. Peter*s Hospital, Chertsey, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared in order to minimize the risk that individual patients could be reidentified, given that there are limited numbers of study participants at each study site per year.

DOCUMENTS (2):
  • Study Protocol (2020-04-08): https://cdn.clinicaltrials.gov/large-docs/19/NCT04506619/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-09): https://cdn.clinicaltrials.gov/large-docs/19/NCT04506619/SAP_001.pdf